CLINICAL TRIAL: NCT06501027
Title: The Effect of Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation on Heart Rate Variability, Psychological Resilience, and Sleep Quality in Earthquake Survivors
Brief Title: Mindfulness-Based Self-Compassion and Vagal Nerve Stimulation on Heart Rate Variability, Psychological Resilience, and Sleep Quality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/07-1075
Record Dates: First submitted 2024-06-04; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Heart Rate Variability; Psychological Resilience; Sleep Quality
Keywords: Mindfulness-Based Self-Compassion Intervention; Vagal Nerve Stimulation; earthquake victims
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Self-Compassion and vagal nerve stimulation (Experimental): Mindfulness-Based Self-Compassion and vagal nerve stimulation were administered to the Intervention I group. Mindfulness-Based Self-Compassion intervention is a manualized course that includes meditation, relaxing movement, and breathing. A certified Mindfulness-Based Self-Compassion instructor will teach the courses in a group-based format for 90 minute sessions, once per week for three weeks.
  Vagal nerve stimulation was administered to all participants in both groups using the on-invasive Auricular Vagus Nerve Stimulation device. The stimulation was biphasic, with a frequency of 10 Hz and a pulse width of 300 μs in Modulation mode. Current intensity was adjusted by attaching the device to the participant's right or left ears, ensuring that they felt the current comfortably, and maintaining a constant level. Stimulation sessions occurred every 3 weeks, with non-invasive auricular vagus nerve stimulation applied for 20 minutes per session over a period of 3 days.
  Interventions: Behavioral: Mindfulness Based Self Compassion
- Vagal nerve stimulation (Experimental): Only vagal nerve stimulation was administered to the Intervention II group. Vagal nerve stimulation was administered to all participants in both groups using the Non-invasive Auricular Vagus Nerve Stimulation device. The stimulation was biphasic, with a frequency of 10 Hz and a pulse width of 300 μs in Modulation mode. Current intensity was adjusted by attaching the device to the participant's right or left ears, ensuring that they felt the current comfortably, and maintaining a constant level. Stimulation sessions occurred every 3 weeks, with non-invasive auricular vagus nerve stimulation applied for 20 minutes per session over a period of 3 days.
  Interventions: Behavioral: Mindfulness Based Self Compassion

INTERVENTIONS:
Behavioral: Mindfulness Based Self Compassion — The intervention has its roots in meditations and yoga practices. However, it is independent of religious purpose or affiliation.The weekly sessions include a range of mental and bodily practices, including awareness of

SUMMARY:
This study was conducted to determine the effects of a mindfulness-based self-compassion intervention and vagal nerve stimulation on heart rate variability, psychological resilience, and sleep quality in earthquake victims.

Design: "The study was designed as a randomized experimental research, where pre- and post-intervention measurements were administered to Intervention I and Intervention II groups."

DETAILED DESCRIPTION:
Hypotheses

H1: The post-intervention sleep quality scores of earthquake victims in the intervention group, who received Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation, will be higher than their scores before the intervention.

H2: The Psychological Resilience Scale scores of earthquake victims in the intervention group, who received Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation, will be higher post-intervention compared to pre-intervention.

H3: The post-intervention heart rate variability of earthquake victims in the Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation intervention group will be higher than their pre-intervention levels.

H4: The earthquake victims in the Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation intervention group will exhibit higher post-intervention sleep quality scores compared to those in the Vagal Nerve Stimulation-only group.

H5: Earthquake victims in the intervention group receiving Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation will demonstrate higher Psychological Resilience Scale scores post-intervention compared to those in the group receiving only Vagal Nerve Stimulation.

H6: Earthquake victims in the intervention group receiving Mindfulness-Based Self-Compassion Intervention and Vagal Nerve Stimulation will show higher post-intervention heart rate variability compared to those in the group receiving only Vagal Nerve Stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 35,
* who have been exposed to an earthquake and have relocated to Istanbul,
* who are accessing psychological first aid information channels.

Exclusion Criteria:

* Individuals with a psychiatric diagnosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-07-12 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | up to 4 weeks
  Heart Rate Variability (HRV) refers to the variation in the time interval between heartbeats. It is a measure of the slight differences in timing between successive heartbeats, often measured in milliseconds. HRV is regulated by the autonomic nervous system, which controls involuntary bodily functions, including heart rate.

SECONDARY OUTCOMES:
Psychological Resilience | up to 4 weeks
  Psychological Resilience Scale for Adults: The scale consists of 33 items; it includes 6 sub-dimensions: The structural style (3,9,15,21) and perception of future (2,8,14,20) subdimensions were measured by 4 items each, the family cohesion (5,11,17,23,26,32), perception of self (1,7,13,19,28,31,), and social competence (4,10,16,22,25,29) subdimensions were measured by 6 items each, and the social resources (6,12,18,24,27,30,33) sub-dimension was measured by 7 items. The score that can be obtained from the scale varies from 33 to 165.
pittsburgh sleep quality index | up to 4 weeks
  It's a self-rated questionnaire that assesses sleep quality and disorders over a one-month period. Seven "component" scores are derived from nineteen separate items. These components include: a) subjective sleep quality, b) sleep latency, c) sleep duration, d) habitual sleep efficiency, e) sleep disorders, f) use of sleeping pills, and g) daytime dysfunction. The sum of these seven component scores yields the index score, with a total score ranging between 0 and 21. A pittsburgh sleep quality index total score of five or higher indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Bat Tonkuş, Dr., Study Chair — İstanbul Yeni Yüzyıl Üniversitesi

IPD SHARING:
Plan to Share IPD: No